CLINICAL TRIAL: NCT07062848
Title: The Transthyretin Amyloid Cardiomyopathy Early Detection With Artificial Intelligence (TRACE-AI) Network Study
Brief Title: An Observational Study Using Artificial Intelligence (AI) Algorithms on Electrocardiography (ECG), Point-of-care Ultrasound (POCUS), and Transthoracic Echocardiophy (TTE) to Estimate the Under-diagnosis of Transthyretin Amyloid Cardiomyopathy (ATTR-CM) Across a Diverse Range of US Health Systems.
Acronym: TRACE Network
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Bridgebio Pharma, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000039184
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Transthyretin (TTR) Amyloid Cardiomyopathy
Keywords: artificial intelligence; AI-ECG; AI-Echo; cardiac amyloidosis; transthyretin amyloid cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: AI Toolkit for ATTR-CM Diagnosis — An artificial intelligence (AI) toolkit of algorithms that detect ATTR-CM on electrocardiography (ECG), point-of-care ultrasound (POCUS), and transthoracic echocardiography (TTE)

SUMMARY:
This is a multi-center, observational study with the overall objective to examine the scale of under-diagnosis for transthyretin amyloid cardiomyopathy (ATTR-CM) across a broad range of diverse health systems in the US using a fully federated deployment of an artificial intelligence (AI) toolkit of algorithms that detect ATTR-CM on electrocardiography (ECG), point-of-care ultrasound (POCUS), and transthoracic echocardiography (TTE).

ELIGIBILITY:
Broad inclusion and exclusion criteria across all 3 objectives:

Inclusion Criteria:

* Age 50-95
* At least one retrievable ECG and/or 2D echo file (DICOM or equivalent video file) from EHR.

Exclusion Criteria:

* Unavailable key demographics (age, gender, race, ethnicity)
* Individuals who have opted out of research studies

Objective-specific inclusion and exclusion criteria:

Primary Objective:

Additional exclusion criteria:

* For subgroup analyses: when evaluating the prevalence of probable ATTR-CM status across demographic groups, we will exclude those with missing baseline demographic information (age, sex, race, geographic region).

Secondary Objective 1:

Additional inclusion criteria:

* 'Cases': ATTR-CM diagnosis defined by ICD-10 codes (Table 1) OR abnormal bone scintigraphy testing consistent with ATTR-CM OR treatment with an approved transthyretin stabilizer or other ATTR-CM-specific therapy
* 'Controls': any individuals not meeting the case definition. In these participants, we will consider all eligible ECG, POCUS, or TTE studies performed up to 12 months before diagnosis (first date of ICD code appearance, abnormal bone scintigraphy or treatment onset, whichever happened first) and any time after. 'Controls' will be drawn from ECGs, POCUS, or TTE studies performed in individuals not meeting the 'case' criteria above, including individuals who have never undergone dedicating testing or those who underwent e.g., bone scintigraphy, but with negative (or equivocal) findings.

Secondary Objective 2:

Additional inclusion criteria:

* Having at least two years of follow-up time between the index test (ECG, POCUS, or TTE) and the date of analysis.
* Having at least one healthcare encounter every two years across care settings from their first entry into the cohort through death or end of the follow-up period.

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include US adults ages 50-95 with at least one retrievable ECG and/or 2D echo file from HER.
Sampling Method: Non-Probability Sample
Enrollment: 1500000 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To describe the prevalence of probable AI-defined ATTR-CM in defined cohorts of individuals who have undergone standard cardiovascular investigations across a diverse network of US-based health care delivery systems | At enrollment

SECONDARY OUTCOMES:
Validate the diagnostic performance of AI-enabled ECG, POCUS, and TTE algorithms for ATTR-CM | At enrollment
To examine the association between the AI-defined probability of ATTR-CM and the incidence of adverse cardiovascular events | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Rohan Khera, MD, MS, Principal Investigator — Yale University
Locations (11):
- United States (11):
  - University of California - San Francisco (UCSF) Health, San Francisco, California
  - Yale New Haven Health System, New Haven, Connecticut
  - Henry Ford Health, Detroit, Michigan
  - Mount Sinai, New York, New York
  - Duke Health, Durham, North Carolina
  - Providence Health, Tigard, Oregon
  - Medical University of South Carolina (MUSC) Health, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Houstin Methodist, Houston, Texas
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - University of Washington Medicine, Seattle, Washington